CLINICAL TRIAL: NCT02125955
Title: Effect of Prebiotic Intake on Adiposity, Satiety and Gut Microbiota in Overweight and Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Children's Hospital (Other)
Responsible Party: Principal Investigator, Dr. Raylene Reimer, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UC-1026386
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Overweight; Obesity
Keywords: Pediatric; Overweight; Obesity; Gut microbiota; Adiposity; Prebiotic; Dietary fiber
MeSH Terms: conditions — Overweight; Obesity | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prebiotic fiber (Experimental): The intervention group will consume an 8 gram dose of prebiotic fiber one time per day approximately 30 minutes prior to their evening meal.
  Interventions: Dietary Supplement: Prebiotic fiber
- Placebo (Placebo Comparator): The placebo group will consume an isocaloric dose of placebo (maltodextrin; 3.3 grams) one time per day approximately 30 minutes prior to their evening meal.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic fiber — Dissolved in water.
  Other Names: Synergy 1 (oligofructose enriched inulin)
  Arms: Prebiotic fiber
Dietary Supplement: Placebo — Dissolved in water
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
Currently, over one third of Canadian children and youth aged five to seventeen are overweight or obese. Childhood obesity leads to increased risks of co-morbidities such as type 2 diabetes, fatty liver disease, cardiovascular disease and certain types of cancers. Changes in the food supply have been linked to obesity and include a decrease in the intake of dietary fiber. Prebiotic fibers are a group of non-digestible carbohydrates that modulate the composition and actions of the gut microbiota and have been shown to reduce body fat and energy intake in overweight and obese adults. The investigators hypothesis is that prebiotic fiber intake in overweight and obese children will similarly result in improvements in body composition and reduced energy intake.

DETAILED DESCRIPTION:
Obesity in the pediatric population is a primary public health concern given that overweight and obesity in childhood continues into adulthood. Consumption of high-fat, calorie-dense diets do not provide individuals with the suggested daily intake of many important nutrients. This is especially true for dietary fiber which has positive health benefits such as roles in weight management. A form of dietary fiber with links to obesity treatment/prevention is prebiotic fiber. In the gut, there are many bacteria which have been shown to affect a person's health depending on the type and number of each type of bacteria. The role of prebiotic fiber is to increase the number of beneficial bacteria which in turn promotes health. Studies in humans have shown that prebiotic fiber is effective at reducing body fat and food intake in overweight and obese adults. The aim of this study is to see if prebiotic fiber can provide the same benefits to overweight and obese children. Since weight management becomes increasingly difficult as a person ages, treatments that promote weight maintenance at an early age are critically needed.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls between the ages of 7-12 years old
* BMI percentiles >85th percentile for their age and sex
* Tanner stage of ≤ 3, girls premenarche

Exclusion Criteria:

* Tanner stage of >3 or girls postmenarchal
* Use of antibiotics up to 3 months prior to study
* Regular prebiotic supplement and/or probiotic supplement use
* Subjects unable to provide consent (parental) or assent (child)

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Body fat | 16 weeks
  Change in baseline fat mass at 16 weeks. Measured by dual energy x-ray absorptiometry.

SECONDARY OUTCOMES:
Appetite regulation | 16 weeks
  Change in baseline appetite at 16 weeks. Subjective appetite assessed with visual analog scales and eating behavior questionnaire. Objective measures include a weighed breakfast buffet, weighted 3-day food records and serum satiety hormone levels.

OTHER OUTCOMES:
Gut microbiota | 16 weeks
  Change in baseline gut microbiota at 16 weeks.
Serum lipids | 16 weeks
  Change in baseline serum lipids at 16 weeks.
Serum glucose and insulin | 16 weeks
  Change in baseline glucose and insulin at 16 weeks.
Inflammatory markers | 16 weeks
  Change in serum inflammatory markers at 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Raylene A Reimer, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Nicolucci AC, Hume MP, Martinez I, Mayengbam S, Walter J, Reimer RA. Prebiotics Reduce Body Fat and Alter Intestinal Microbiota in Children Who Are Overweight or With Obesity. Gastroenterology. 2017 Sep;153(3):711-722. doi: 10.1053/j.gastro.2017.05.055. Epub 2017 Jun 5. PMID 28596023
- [Result] Hume MP, Nicolucci AC, Reimer RA. Prebiotic supplementation improves appetite control in children with overweight and obesity: a randomized controlled trial. Am J Clin Nutr. 2017 Apr;105(4):790-799. doi: 10.3945/ajcn.116.140947. Epub 2017 Feb 22. PMID 28228425